CLINICAL TRIAL: NCT01983332
Title: Impact of the Introduction of Model of Human Occupation (MOHO) on Clinical Reasoning in Therapists Working With Clients in the Cancer Population
Brief Title: Impact of MOHO on Therapists Working With Clients in Cancer Population
Acronym: MDACC-MOHO
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Patricia Bowyer, Patricia Bowyer, EdD, MS, OTR, FAOTA, Texas Woman's University
Other Study IDs: 17075
Record Dates: First submitted 2013-07-05; First posted 2013-11-14 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Cancer
Keywords: MDACC; MOHO
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- occupational therapists: Occupational Therapists

SUMMARY:
The purpose of this study is to examine the impact of an introduction to the occupation-based theory (MOHO) on the clinical reasoning of therapists working with cancer clients.

DETAILED DESCRIPTION:
The study will occur at MDACC, a comprehensive cancer center in the Texas Medical Center (TMC) in Houston. The center is the largest freestanding comprehensive cancer center in the world. The facility provides inpatient and outpatient services and supports research and education.

The facility has more than 50 buildings in the greater Houston area and in central Texas. The setting for this study will be the rehabilitation services area on the main campus in the TMC.

There are private offices, conference rooms and treatment areas where video chats and monthly meetings will occur.

The study is projected to occur over a one year period. Sessions will be videotaped (video chats - initial and follow ups and monthly group meetings) for further review. Analysis of the tapes will provide data for further research and education presentations. Sessions will also be audiotaped and transcribed for further review and data analysis purposes. Neither the videotapes nor audiotapes will be shared with anyone at the facility or any uninvolved parties. Audiotapes and videotapes will be stored in locked file cabinets and password protected computers will be used to view and analyze the audio and video tapes. Only the research team will have access to the stored data locked in the file cabinet.

ELIGIBILITY:
Inclusion Criteria:

No training in MOHO constructs,English speaking.

Exclusion Criteria:

Training in using MOHO concepts in practice, highly skilled in use of MOHO, and non-English speaking. If a therapist is skilled and knowledgeable of the constructs of MOHO, there will be no way to determine if introduction of the model has impacted a therapist's clinical reasoning. All the materials used for the study will be in English and analysis of data will be conducted by English speaking individuals, therefore the study participants must speak English.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be outpatient-focused therapists working within the MD Anderson Cancer Center. Participants must have worked in this setting for at least 90 days before the study begins and will self-select to participate in the study. Recruitment of therapists at the MDACC will involve an introduction of the study by an onsite collaborator. The onsite collaborator will gather the names of individuals interested in participating in the study. Then, an onsite collaborator and PI will work together to determine if the therapists meet the inclusion criteria for the study. Once the therapists are determined to meet inclusion criteria, an invitation for participation will be extended by an onsite collaborator.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Interviews and training sessions-observational analysis of video taped sessions | 30 1/2 hours over course of year
  The study will begin with a video chat (20-30 minutes) to attain a baseline of participants understanding of MOHO. An initial video chat interview guide (Appendix B) will be used to facilitate the chat session and a training session on MOHO concepts (4-8 hours) will also be held (Appendix F). The training session is a 6 part overview of the MOHO framework. All following video chats will be conducted using the follow up video chat interview guide (Appendix C). There will be 8 follow up video chat sessions (20-30 minutes) occurring every 6 weeks after the initial training session on MOHO concepts. Video chat sessions will be facilitated by a research team member. There will be 12 monthly group meetings (60-90 minutes) with all participants to allow a time to discuss use of MOHO in practice and troubleshoot issues and offer support in a formal manner. The monthly group meeting will be facilitated by the PI and/or an onsite collaborator. The maximum possible time commitment stands at 1830

SECONDARY OUTCOMES:
Observational data analysis-theme sorting until saturation reached | 1 year
  This is a qualitative study and data will be analyzed using theme sorting until commonn themes are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bowyer, EdD,MS,OTR, Principal Investigator — Texas Woman's University
Locations (2):
- United States (2):
  - M.D. Anderson Cancer Center, Houston, Texas
  - Texas Woman's University, Houston, Texas